CLINICAL TRIAL: NCT03315429
Title: Unmasking the Dynamic Component in Functional Mitral Regurgitation in Chronic Heart Failure
Acronym: ALLEGRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Georg Goliasch, Asc.Prof. Priv.Doz. Dr., PhD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1590/2017
Record Dates: First submitted 2017-10-10; First posted 2017-10-20 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stress testing arm (Other): Stress testing of patients with functional mitral regurgitation.
  Interventions: Diagnostic Test: stress echocardiography

INTERVENTIONS:
Diagnostic Test: stress echocardiography — stress testing of patients with functional mitral regurgitation

SUMMARY:
Background:

Chronic heart failure (HF) is frequently accompanied by functional mitral regurgitation (FMR) caused by left ventricular (LV) remodeling and subsequent papillary muscle displacement resulting in mitral valve (MV) leaflet tethering, dilatation and flattening of the mitral annulus and reduced closing forces. Up to moderate FMR affects the majority of patients with systolic heart failure - roughly 80% - still independently increasing mortality. Every fifth patient with chronic heart failure experiences a progression of FMR during the first three years of follow up despite guideline directed heart failure therapy, which is independently associated with a poor prognosis. Furthermore, MR is well known to have a strong dynamic component not only during the cardiac cycle at rest and with exercise.

Aims of the study:

The investigators therefore aim to assess whether stress tests in patients with functional mitral regurgitation unmasks significant dynamic mitral regurgitation or might aid to identify patients at risk of FMR progression in patients with functional mitral regurgitation in heart failure with reduced ejection fraction (HFrEF) under guideline directed medical therapy.

Study design:

The investigators will prospectively perform stress tests in all patients with non-severe FMR that are routinely seen in the heart failure outpatient clinic.

Study patients:

Patients with stable chronic heart failure on optimal medical therapy, who undergo routine ambulatory clinical control visits in the heart failure outpatient ward of the Medical University of Vienna, will be included in the present study. A written informed consent will be obtained before inclusion. Inclusion criteria will be a non-severe FMR, an age of at least 18 years and stable heart failure related medical therapy in the last 3 months.

Methods:

All patients that are willing to participate will undergo stress testing (i.e. volume challenge and low dose dobutamine stress) to determine whether patients display severe dynamic FMR under stress conditions. Within the registry patients will be followed-up during routine ambulatory visits for three years. Patients with severe dynamic functional mitral regurgitation will be compared to patients without severe dynamic FMR. Record of clinical events during the FUP will be performed. Routine laboratory parameters, have been measured at inclusion. Additionally, neurohormone patterns will be measured at baseline and at peak stress.

Sample size:

Expecting a prevalence of severe dynamic FMR of 20%, the investigators would include a total of 150 chronic heart failure patients taking also into account a study-dropouts of 20% ( loss of follow-up and mortality).

ELIGIBILITY:
Inclusion Criteria:

* non-severe FMR,
* age of at least 18 years,
* stable heart failure related medical therapy in the last 3 months.

Exclusion criteria

* non-willing to participate
* myocardial infarction,
* cardiac decompensation within the last 3 months,
* pregnancy,
* life expectancy of less than 1 year for non cardiac reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of severe dynamic FMR under stressed conditions | 3 years

SECONDARY OUTCOMES:
Identification of a relationship between dynamic FMR (defined as advance of at least one grade in severity with transition to at least moderate during stress) and FMR progression during rest within the 3 year follow-up period. | 3 years
correlation of the prevalence of dynamic FMR with the dynamic levels of neurohormones | 3 years
Establishment of an association between dynamic FMR and outcome (combined measure consisting of hospitalization for heart failure and/or death) during the follow-up period | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria